CLINICAL TRIAL: NCT01263704
Title: A Phase II, Multicenter, Single Arm Study to Determine the Efficacy and Safety of Low Dose Fludarabine and Cyclophosphamide Combined With Standard Dose Rituximab as Primary Therapy in Elderly Untreated Patients (>/=65 Years Old) With Chronic Lymphocytic Leukemia
Brief Title: A Study of MabThera/Rituxan (Rituximab) in Combination With Fludarabine And Cyclophosphamide as Primary Therapy in Elderly Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25464
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rituximab plus Fludarabine and Cyclophosphamide (Experimental): Elderly participants with chronic lymphocytic leukemia (CLL) will receive combination treatment with low-dose fludarabine and cyclophosphamide combined with standard-dose of rituximab for 6 months. Treatment is followed by a follow up period of 36 months.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — 150 milligrams per square meter (mg/m^2) intravenously (IV) on Days 1-3 of each 28-day cycle for 6 cycles
Drug: Fludarabine — 12.5 mg/m^2 IV on Days 1-3 of every 28-day cycle for 6 cycles
Drug: Rituximab — 375 mg/m^2 IV Day 0 of Cycle 1, 500 mg/m^2 IV Day 1 of Cycles 2-6. Each cycle was 28 days.
  Other Names: MabThera/Rituxan

SUMMARY:
This single arm, open-label study will assess the safety and efficacy of low dose fludarabine and cyclophosphamide in combination with standard dose MabThera/Rituxan (rituximab) as primary therapy in elderly patients (>/= 65 years) with chronic lymphocytic leukemia. Patients will receive six 28-day cycles of treatment with Mabthera/Rituxan (375 mg/m2 intravenously [iv] Day 0 of cycle 1, 500 mg/m2 iv Day 1 of cycles 2-6), fludarabine (12.5 mg/m2/d iv Days 1-3, cycles 1-6) and cyclophosphamide (150 mg/m2/d iv Days 1-3, cycles 1-6). Anticipated time on study treatment is 6 months, with a 30-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 65 years of age
* Previously untreated B-cell chronic lymphocytic leukemia (CLL)
* Binet stage C or active Binet stage A and B disease

Exclusion Criteria:

* Prior treatment for CLL
* CLL with transformation (Richter's syndrome)
* Suspected or known central nervous system (CNS) involvement of CLL
* Impaired renal or hepatic function
* Human Immunodeficiency Virus (HIV) positivity, active hepatitis B/C or Hepatitis B Virus (HBV) surface antigen positive, or any active or uncontrolled infections
* Patients with anti-HBV core antibodies (past infection with HBV) but who are negative for Hepatitis B Virus Surface Antigen (HBVsAg) (either anti-HBS Ab positive or negative) and are positive for HBV- Deoxyribonucleic acid (DNA) by Polymerase chain reaction (PCR) analysis
* Concomitant diseases requiring chronic steroid administration
* Active second malignancy within the 2 years prior to study (except for non-melanoma skin cancer and in situ cervix or breast or prostate carcinoma)
* Eastern Cooperative Oncology Group (ECOG) performance status >/= 3

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07-17 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Israel (12):
  - Haemek Medical Center; Hematology Department, Afula
  - Soroka Medical Center; Hematology Deptartment, Beersheba
  - Rambam Medical Center; Heamatology & Bone Marrow Transplantation, Haifa
  - Bnei-Zion Medical Center; Hematology Dept, Haifa
  - Shaare Zedek Medical Center; Hematology Dept., Jerusalem
  - Hadassah Ein Karem Hospital; Haematology, Jerusalem
  - Meir Medical Center; Internal Dept A, Kfar Saba
  - Western Galilee Hospital - Nahariya, Nahariya
  - Beilinson Medical Center; Haematology, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - ASSAF Harofe; Department of Hematology, Rishon LeZiyyon
  - Ichilov Sourasky Medical Center; Heamatology, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab Plus Fludarabine and Cyclophosphamide: Elderly participants with chronic lymphocytic leukemia (CLL) received combination treatment with low-dose fludarabine and cyclophosphamide combined with standard-dose of rituximab for 6 months. Treatment was followed by a follow up period of 36 months.
Period: Overall Study
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Started | 42
Completed | 13
Not Completed | 29
Not completed — Progressive disease | 18
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Patient withdrew consent | 2
Not completed — Eligibility criteria not fulfilled | 1
Not completed — Lost to Follow-up | 1
Not completed — Colon metastases | 1
Not completed — Principal Investigator (PI) decision | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all enrolled participants.
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate was defined as the percentage of participants with a complete response (CR) or a partial response (PR) according to National Cancer Institute - Working Group [NCI-WG] guidelines. CR: no clonal B lymphocytes in peripheral blood, no significant lymphadenopathy, liver and spleen normal size, no disease symptoms, blood counts: absolute neutrophil count (ANC) >1,500/microliter (mcL), platelets > 100,000/mcL, hemoglobin > 11.0 grams/deciliter (g/dL), normocellular bone marrow. PR: >/= 50% decrease in clonal B lymphocyte count, >/= 50% reduction in lymphadenopathy, >/= 50% reduction of liver or spleen enlargement and ANC >1,500/mcL, platelets > 100,000/mcL, hemoglobin > 11.0 g/dL OR >/= 50% increase in ANC, platelets or hemoglobin.
Time Frame: Up to 42 months
Population: Efficacy analysis population included all participants who received rituximab during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 40
percentage of participants | 67.5 [50.9 to 81.4]

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Preexisting conditions which worsen during a study are also considered as adverse events. An SAE is any experience that suggests a significant hazard, contraindication, side effect, or precaution, and fulfills any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here.
Time Frame: Up to 53 months
Population: The safety population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 42
percentage of participants
  AEs | 97.6
  SAEs | 45.2

3. Secondary Outcome: Percentage of Participants With Neutropenic Fever, Infection, >/= Grade 3 Drug-Related Neutropenia, >/= Grade 3 Drug-Related Thrombocytopenia, Hospitalizations
Time Frame: Up to 53 months
Population: The safety population included all enrolled participants.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 42
percentage of participants
  Infection | 47.6
  Neutropenic fever | 14.3
  ≥ Grade 3 drug-related neutropenia | 47.6
  ≥ Grade 3 drug-related thrombocytopenia | 11.9
  Hospitalization | 19.1

4. Secondary Outcome: Hospitalization Days
Time Frame: Up to 53 months
Population: The safety population included all enrolled participants.
Measure: Median (Full Range); unit: days
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 42
days | 8 [2 to 13]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval from the first study drug treatment day to the first sign of disease progression according to NCI-WG guidelines. Progressive disease (PD): Any new lesion, any disease symptoms, >/=50% increase in lymphadenopathy, splenomegaly, hepatomegaly, >/= 50% increase in the number of circulating clonal B lymphocytes, decrease of hemoglobin levels by > 2.0 g/dL, >/= 50% decrease of platelet counts, increase of lymphocytes in bone marrow to more than 30% from normal.
Time Frame: Up to 53 months
Population: Efficacy analysis population included all participants who received rituximab during the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 40
months | 36.1 [27.3 to 48.1]

6. Secondary Outcome: Quality of Life (QoL): Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Questionnaire
Description: The FACIT-F questionnaire consists of 13 questions with a total score range of 0 to 52 with 0 indicating a better outcome and 52 indicating a worse outcome.
Time Frame: [Visit 1 (Screening, Week 0), at Visits 11 (Week 45) and 14 (Week 80) and at the end of the study (Month 42)]
Population: Efficacy analysis population included all participants who received rituximab during the study. Participants from the efficacy analysis population, who completed the FACIT-F questionnaire at any time point during the study, were analyzed as indicated at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
Number analyzed (Participants) | 40
score on a scale
  Visit 1 (Screening, Week 0): number analyzed (Participants) | 30
  Visit 1 (Screening, Week 0) | 36.1 (11.1)
  Visit 11 (Week 45): number analyzed (Participants) | 23
  Visit 11 (Week 45) | 39.4 (9.2)
  Visit 14 (Week 80): number analyzed (Participants) | 13
  Visit 14 (Week 80) | 40.2 (10.1)
  End of the Study (Month 42): number analyzed (Participants) | 3
  End of the Study (Month 42) | 47.0 (1.0)

ADVERSE EVENTS:
Time Frame: Up to 53 months
Description: The safety population included all enrolled participants.
Arm/Group | Rituximab Plus Fludarabine and Cyclophosphamide
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 19/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Fludarabine and Cyclophosphamide (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diabetes mellitus (Endocrine disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Pyrexia (General disorders) | 3
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia bacterial (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Subacute endocarditis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Delirium (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab Plus Fludarabine and Cyclophosphamide (N=42)
Anemia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 8
Chills (General disorders) | 4
Fatigue (General disorders) | 4
Infusion related reaction (General disorders) | 5
Edema peripheral (General disorders) | 3
Pyrexia (General disorders) | 4
Pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Neutrophil count decreased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT01263704/Prot_SAP_000.pdf